CLINICAL TRIAL: NCT02720224
Title: An Open-Label, Single Dose Study Designed to Assess the Mass Balance Recovery, Metabolite Profiles and Metabolite Identification of [14C]-Estetrol in Healthy Female Volunteers
Brief Title: Study Conducted to Further Understand the Elimination Pathways, Metabolite Profile and PK Profile of 14C-estetrol
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Estetra (Industry)
Collaborators: Quotient Clinical (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: MIT -Es0001-C105; 2014-000622-38 (EudraCT Number)
Record Dates: First submitted 2016-01-08; First posted 2016-03-25 (Estimated); Results first posted 2018-12-10 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2016-01

CONDITIONS: Contraception; Menopause
MeSH Terms: interventions — Estetrol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Estetrol (Experimental): A single oral dose of 15 mg carbon 14 labelled estetrol ([14C]-estetrol), containing approximately 2.8 MBq (76 µCi) 14C
  Interventions: Drug: Estetrol

INTERVENTIONS:
Drug: Estetrol — 15 mg [14C]-estetrol containing approximately 2.8 MBq (76 μCi) 14C
  Other Names: E4

SUMMARY:
This study is being conducted to further understand the elimination pathways, metabolite profile and pharmacokinetic (PK) profile of carbon 14 labelled estetrol ([14C] estetrol).

DETAILED DESCRIPTION:
This will be an open-label, non-randomised, single dose study in healthy female volunteers of non-child bearing potential.

Subjects will be screened for eligibility to participate in the study up to 28 days before dosing. The study will be executed in a single group, 6 subjects will be enrolled and dosed with a single oral dose of carbon 14 labelled estetrol. Subjects will be admitted to the clinical unit on the morning prior to study drug administration (Day -1). Dosing will take place on the morning of Day 1 after an overnight fast (approximately 10 h).

Subjects will be resident in the clinic up to 240 h after dosing during which plasma, blood, urine and faeces samples will be collected. It is planned that subjects will be released as a group when all subjects have achieved a mass balance cumulative recovery of >90% or if a mean of <1% of the dose administered has been collected in urine and faeces within 2 separate, consecutive 24 h periods. In this case, collection of all samples (blood, urine and faeces) will be stopped and the subjects will undergo discharge assessments. If this criterion has not been met by all subjects on Day 11, home collections of urine and faeces may be requested at the discretion of the investigator for individual subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy females of non-child bearing potential, i.e. surgically sterilised or post menopausal subjects. Postmenopausal status will be defined by an absence of menses for a minimum of 12 months and confirmed by a FSH result ≥30 IU/ml
2. Negative pregnancy test at screening and Day -1
3. 30 to 65 years of age inclusive
4. Body mass index between ≥18.0 and ≤30.0 kg/m2
5. Must be willing and able to communicate and participate in the whole study
6. Must provide written informed consent
7. Must have regular bowel movements (i.e. average stool production of ≥1 and ≤3 stools per day)Must agree to use an adequate method of contraception

Exclusion Criteria:

1. Participation in a clinical research study within the previous 3 months
2. Subjects who are study site employees, or immediate family members of a study site or sponsor employee
3. Subjects who have previously been enrolled in this study
4. History of any drug or alcohol abuse in the past 2 years
5. Regular alcohol consumption i.e. >14 units per week (1 unit = ½ pint beer, 25 ml of 40% spirit or a 125 ml glass of wine)
6. Current smokers and those who have smoked within the last 12 months. A breath carbon monoxide reading of greater than 10 ppm at screening
7. Females who are pregnant or lactating
8. Radiation exposure, including that from the present study, excluding background radiation but including diagnostic x-rays and other medical exposures, exceeding 5 mSv in the last 12 months or 10 mSv in the last 5 years. No occupationally exposed worker, as defined in the Ionising Radiation Regulations 1999, shall participate in the study
9. Subjects who do not have suitable veins for multiple venepunctures/cannulation as assessed at screening
10. Clinically significant abnormal biochemistry, haematology or urinalysis as judged by the investigator
11. Positive drugs of abuse test result
12. Positive hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV Ab) or human immunodeficiency virus (HIV) results
13. History or presence of clinically significant cardiovascular, renal, hepatic, chronic respiratory or gastrointestinal disease as judged by the investigator
14. Serious adverse reaction or serious hypersensitivity to any drug or the formulation excipients
15. Presence or history of clinically significant allergy requiring treatment, as judged by the investigator. Hayfever is allowed unless it is active
16. Donation or loss of greater than 400 ml of blood within the previous 3 months
17. Subjects who are taking, or have taken, any prescribed medications in the 28 days before IMP administration (exceptions may apply on a case by case basis provided they are considered not to interfere with the objectives of the study as agreed by the PI or delegate and sponsor's medical monitor), or over-the-counter drug or herbal remedies in the 14 days before IMP administration. If needed (i.e. an incidental and limited need) ibuprofen is acceptable as analgesic treatment, but must be documented in the (Case Report Form) CRF. Use of paracetamol is forbidden during the entire study
18. Subjects who are not in euthyroid condition (thyroid-stimulating hormone [TSH] and free thyroxine [fT4] within the normal reference range)
19. Any history of suspected malignancy with the exception of basal cell (excluded if within the prior 2 years) or squamous cell (excluded if within the prior one year) carcinoma of the skin
20. History or presence of prolonged QT interval corrected by Bazett's formula or any other clinically significant ECG abnormalities as judged by the investigator based on 12-lead ECG readings at screening
21. Subjects with abnormal supine blood pressure at screening: at least 2 readings of systolic blood pressure greater than 140 mmHg or lower than 90 mmHg, and/or diastolic blood pressure of more than 90 mmHg or lower than 50 mmHg after minimum intervals of 5 min
22. Any surgical or medical condition which might significantly alter the absorption, distribution, metabolism, or excretion of drugs, or which may jeopardize the subject in case of participation in the study. The investigator should make this determination in consideration of the subject's medical history and/or clinical or laboratory evidence of any of the following:

    * History or symptoms of inflammatory bowel disease, gastritis, ulcers, gastrointestinal or rectal bleeding,
    * History of major gastrointestinal tract surgery (subjects who have had an appendectomy are acceptable for inclusion),
    * History or presence of pancreatic injury or pancreatitis,
    * History or presence of impaired hepatic function,
    * History or presence of liver disease or liver injury as indicated by abnormal liver function tests such as aspartate aminotransferase (AST), alanine aminotransferase (ALT), gamma-glutamyl transferase (GGT), alkaline phosphatase (ALP), or total serum bilirubin. Any single parameter elevated ≥1.5 fold upper limit of normal should be re-checked once prior to enrolment/randomisation (subject who have had a cholecystectomy are acceptable for inclusion if all liver/gallbladder parameters are in the normal range),
    * History or presence of impaired renal function if considered as clinically significant,
    * Abnormal urinary constituents (e.g. albumin if considered as clinically significant).
23. Suspected or current history of gynaecological or breast pathology, including any abnormal Pap smear within the 3 previous years (ASCUS , ASC-H , LGSIL or worse) or history of abnormal mammogram within the 2 previous years
24. Failure to satisfy the investigator of fitness to participate for any other reason

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2016-02; Primary Completion 2016-03 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Litza McKenzie, MBChB, Principal Investigator — Quotient Clinical
Locations (1):
- Quotient Clinical, Ruddington, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Estetrol
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Estetrol
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.8 (3.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 0
Region of Enrollment [Number; unit: participants]
  United Kingdom | 6

OUTCOME MEASURES:

1. Primary Outcome: Mass Balance of Total Radioactivity in Urine
Description: Amount excreted in urine (Ae[urine])
Time Frame: From Day -1 prior study treatment intake to 312 hours post-dose
Population: Mass balance population - n = all subjects who took one dose of study treatment and had evaluable total radioactivity concentration (urinary and faecal) data.
Measure: Mean (Standard Deviation); unit: Cumulative percent excreted (%)
Arm/Group | Estetrol
Number analyzed (Participants) | 6
Cumulative percent excreted (%) | 68.97 (7.30)

2. Primary Outcome: Mass Balance of Total Radioactivity in Faeces:
Description: Amount excreted in faeces (Ae[faeces])
Time Frame: From Day -1 prior study treatment intake to 312 hours post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Cumulative percent excreted (%)
Arm/Group | Estetrol
Number analyzed (Participants) | 6
Cumulative percent excreted (%) | 21.88 (8.29)

3. Secondary Outcome: Maximum Concentration (Cmax) of Total Radioactivity in Plasma
Time Frame: Predose, 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 5, 6, 8, 12, 16, 24, 36, 48, 72, 96, 120, 144, 168, 192, 216, 240 hours post-dose
Population: Pharmacokinetic (PK) population - n = all subjects who took one dose of study treatment and had sufficient quantifiable post-dose plasma concentration for PK parameter estimation.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Estetrol
Number analyzed (Participants) | 6
ng/mL | 231 (29.2)

4. Secondary Outcome: Time to Maximum Concentration (Tmax) of Total Radioactivity in Plasma
Time Frame: as for outcome 3
Population: PK population - n = all subjects who took one dose of study treatment and had sufficient quantifiable post-dose plasma concentration for PK parameter estimation.
Measure: Median (Full Range); unit: hour
Arm/Group | Estetrol
Number analyzed (Participants) | 6
hour | 0.25 [0.25 to 0.50]

5. Secondary Outcome: Area Under the Curve From 0 Time to Last Measurable Concentration [AUC(0-last)] of Total Radioactivity in Plasma
Time Frame: as for outcome 3
Population: PK population - n = all subjects who took one dose of study treatment and had sufficient quantifiable post-dose plasma concentration for PK parameter estimation.
  One subject was excluded from the AUC0-last calculation due to undetectable samples from 4 to 24 hours post E4 dose.
Measure: Median (Full Range); unit: ng*h/mL
Arm/Group | Estetrol
Number analyzed (Participants) | 5
ng*h/mL | 561 [369 to 819]

6. Secondary Outcome: The Elapsed Time (Tlag) of Total Radioactivity in Plasma
Time Frame: as for outcome 3
Population: as for outcome 4
Measure: Median (Full Range); unit: hour
Arm/Group | Estetrol
Number analyzed (Participants) | 6
hour | 0.0 [0.0 to 0.0]

7. Secondary Outcome: Cmax of Estetrol in Plasma
Time Frame: as for outcome 3
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Estetrol
Number analyzed (Participants) | 6
ng/mL | 16.6 (18.7)

8. Secondary Outcome: Tmax of Estetrol in Plasma
Time Frame: as for outcome 3
Population: as for outcome 4
Measure: Median (Full Range); unit: hour
Arm/Group | Estetrol
Number analyzed (Participants) | 6
hour | 0.25 [0.25 to 0.50]

9. Secondary Outcome: AUC(0-last) of Estetrol in Plasma
Time Frame: as for outcome 3
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Estetrol
Number analyzed (Participants) | 6
ng*h/mL | 90.4 (15.4)

10. Secondary Outcome: AUC(0-infinity) of Estetrol in Plasma
Time Frame: as for outcome 3
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Estetrol
Number analyzed (Participants) | 6
ng*h/mL | 92.6 (15.2)

11. Secondary Outcome: Tlag of Estetrol in Plasma
Time Frame: as for outcome 3
Population: as for outcome 4
Measure: Median (Full Range); unit: hour
Arm/Group | Estetrol
Number analyzed (Participants) | 6
hour | 0.0 [0.0 to 0.0]

12. Secondary Outcome: Half-life (t1/2) of Estetrol in Plasma
Time Frame: as for outcome 3
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour
Arm/Group | Estetrol
Number analyzed (Participants) | 6
hour | 31.7 (31.8)

13. Secondary Outcome: The Mean Residence Time (MRT) of Estetrol in Plasma
Time Frame: as for outcome 3
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour
Arm/Group | Estetrol
Number analyzed (Participants) | 6
hour | 42.78 (31.0)

14. Secondary Outcome: Cmax of Total Radioactivity in Whole Blood
Time Frame: as for outcome 3
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng eq/mL
Arm/Group | Estetrol
Number analyzed (Participants) | 6
ng eq/mL | 122 (27.6)

15. Secondary Outcome: The Terminal Elimination Rate Constant (Lambda-z) of Estetrol in Plasma
Time Frame: as for outcome 3
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: 1/hour
Arm/Group | Estetrol
Number analyzed (Participants) | 6
1/hour | 0.0218 (31.8)

16. Secondary Outcome: AUC(0-last) of Total Radioactivity in Whole Blood
Time Frame: as for outcome 3
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng eq*h/mL
Arm/Group | Estetrol
Number analyzed (Participants) | 6
ng eq*h/mL | 125 (51.7)

17. Secondary Outcome: Renal Clearance (CLr) for Estetrol
Time Frame: From Day-1 prior study treatment intake to 240 hours post-dose
Population: PK and mass balance populations - n = all subjects who took one dose of study treatment and had sufficient quantifiable post-dose samples (plasma, urinary and faecal) for PK and mass balance parameter estimation.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/min
Arm/Group | Estetrol
Number analyzed (Participants) | 6
mL/min | 8.1 (41.6)

18. Secondary Outcome: Renal Clearance (CLr) for Total Radioactivity
Time Frame: From Day-1 prior study treatment intake to 240 hours post-dose
Population: PK and mass balance populations - n = all subjects who took one dose of study treatment and had sufficient quantifiable post-dose samples (plasma, urinary and faecal) for PK and mass balance parameter estimation.
  One subject was excluded from the CLr analysis due to undetectable PK samples from 4 to 24 hours post E4 dose.
Measure: Geometric Least Squares Mean (Geometric Coefficient of Variation); unit: mL/min
Arm/Group | Estetrol
Number analyzed (Participants) | 5
mL/min | 273 (27.0)

19. Secondary Outcome: Number of Subjects With Adverse Events as a Measure of Safety and Tolerability
Time Frame: From maximum 28 days prior study treatment intake to 240 hours post-dose
Population: Safety population - all subjects who took one dose of study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Estetrol
Number analyzed (Participants) | 6
Participants | 2

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from screening (28 days before dosing) to Day 11 post-dose.
Arm/Group | Estetrol
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 2/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Estetrol (N=6)
BLOOD THYROID STIMULATING HORMONE INCREASED (Investigations) | 1 (1)
NASOPHARYNGITIS (Infections and infestations) | 1 (1)
BLISTER (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes